CLINICAL TRIAL: NCT04331951
Title: Sensitivity of Targeted Biopsy Within Sydney Protocol by Using Narrow Band Imaging for Extensive Gastric Intestinal Metaplasia Diagnosis
Brief Title: Sensitivity of Targeted Biopsy Within Sydney Protocol for GIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principal investigator, King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP016
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Intestinal Metaplasia

STUDY DESIGN:
Masking Description: The pathologists will be blinded for the result of endoscopic finding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted biopsy within Sydney Protocol (Experimental): The patients with history of gastric intestinal metaplasia will be included and using targeted biopsy within Sydney Protocol; both targeted biopsy at suspicious lesions and random biopsy at no suspicious area.
  * All tissues will be sent to immunohistochemistry as a gold standard.
  * Sensitivity, specificity,positive predictive value, negative predictive value, accuracy will be calculated.
  Interventions: Diagnostic Test: Targeted biopsy within Sydney protocol

INTERVENTIONS:
Diagnostic Test: Targeted biopsy within Sydney protocol — Biopsy at suspicious GIM lesions at any area of antrum (both lesser and greater curvature site), body (both lesser and greater curvature site) and incisura. If there is no abnormal mucosa seen at any site, random biopsy will be performed.

SUMMARY:
Sensitivity of Targeted Biopsy Within Sydney Protocol by Using Narrow Band Imaging for Extensive Gastric Intestinal Metaplasia Diagnosis

Objective:

The aim of this study is to evaluate the sensitivity of targeted biopsy within Sydney protocol by using narrow band imaging for Extensive Gastric Intestinal Metaplasia diagnosis

Research design: Diagnosis study

Sample size: 105 cases

Data analysis:

The outcomes will be presented using 2 by 2 tables and if the data are normal distribution the categorical data will be analysed using McNemar's test

DETAILED DESCRIPTION:
Background and Rationale:

Gastric cancer has been in the top-5 of cancer-related death worldwide. Early detection by screening program in high risk patients is very important. If we can detect pre-malignant lesion eg. gastric intestinal metaplasia, we can provide the appropriate surveillance program to those patients. However, the screening protocol for gastric intestinal metaplasia remained unclear. Recently in July 2019, British Society of Gastroenterology published the guideline on the diagnosis and management of patients at risk of gastric adenocarcinoma. The image-enhanced endoscopy (IEE) is recommended as the best modality for assessing gastric intestinal metaplasia. Additionally, they recommended taking biopsy by using Sydney protocol which means taking biopsy at two areas for antrum, two areas for body and one for incisura although they look normal. We aimed to evaluate the sensitivity of this protocol for extensive gastric intestinal metaplasia (GIM) diagnosis in this study.

Methodology:

* All patients with history of GIM will be enrolled and undergone standard with white light esophagogastroduodenoscopy (EGD).
* Those with suspected lesions of GIM will proceed to narrow band imaging (NBI)-mode endoscopy.
* Targeted biopsy will be done at the suspected GIM lesions. Random biopsy will be while will be done if no suspicious GIM lesion seen.

Data collection:

All data will be processed and recorded by one physician.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 year of age
* Suspected GIM by previous tissue pathology
* Able to provide informed consent for participation

Exclusion Criteria:

* Previous gastric surgery including gastrectomy and bypass surgery
* Coagulopathy
* Pregnancy
* Active upper GI bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of targeted biopsy within Sydney protocol by using narrow band imaging for Extensive Gastric Intestinal Metaplasia diagnosis | 4 weeks after completing the enrollment.
  Sensitivity of targeted biopsy within Sydney protocol by using narrow band imaging for Extensive Gastric Intestinal Metaplasia diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand